CLINICAL TRIAL: NCT00887458
Title: A Randomized Phase II Clinical Trial of Two Dose-levels of Itraconazole in Patients With Metastatic Castration-resistant Prostate Cancer
Brief Title: A Two-dose Level Clinical Trial of Itraconazole in Patients With Metastatic Prostate Cancer Who Have Had Disease Progression While on Hormonal Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0932; JHMI-IRB number: NA_00027099
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Results first posted 2014-01-27 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
Keywords: metastatic prostate cancer; castration resistant prostate cancer; rising PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low Dose (Active Comparator): Itraconazole, 200 mg, by mouth, once daily (200 mg total daily dose)
  Interventions: Drug: Itraconazole 200 mg
- High Dose (Active Comparator): Itraconazole, 300 mg, by mouth, twice daily (600 mg total daily dose)
  Interventions: Drug: Itraconazole 300mg

INTERVENTIONS:
Drug: Itraconazole 200 mg — Itraconazole, 200 mg, by mouth, once daily (200 mg total daily dose)
  Arms: Low Dose
Drug: Itraconazole 300mg — Itraconazole, 300 mg, by mouth, twice daily (600 mg total daily dose)
  Arms: High Dose

SUMMARY:
This research is being done to test an investigational drug, called itraconazole, in the treatment of prostate cancer. Itraconazole is approved by the Food and Drug Administration (FDA) for the treatment of various fungal infections such as fingernail/toenail infections and other more serious fungal infections. The word "investigational" means that itraconazole is not approved for use in people with cancer. However, the FDA is allowing the use of itraconazole in this research study. Itraconazole has been shown to have activity against cancer (including prostate cancer) in the laboratory, but has not been tested against cancer in humans.

The purpose of this study is to find out:

* If itraconazole is safe when given at two different doses
* How itraconazole affects prostate specific antigen (PSA): a blood test that measures substances released by prostate cancer
* Whether itraconazole can delay further prostate cancer growth and spread
* How itraconazole affects other markers of prostate cancer

DETAILED DESCRIPTION:
Itraconazole is an oral, generic, and commercially available antifungal drug with a long safety record when used at doses ranging from 200 to 600 mg daily.

Itraconazole has been shown in cellular and animal models to be a potent angiogenesis inhibitor as well as a Hedgehog pathway antagonist; both pathways are considered important in prostate cancer. Itraconazole has not previously been tested as an antineoplastic agent, but given its well-established safety profile, the gap between further preclinical studies and human clinical trials can be narrowed to accelerate development of this agent as a putative anticancer drug. The investigators hypothesize that itraconazole will prevent PSA progression in a significant proportion of men with metastatic CRPC and that it will have an acceptable safety profile at both doses. Itraconazole may ultimately delay the need for chemotherapy in these men.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate adenocarcinoma.
* Presence of distant metastases on bone scan, CT scan, or MRI scan.
* Progression after androgen deprivation (and anti-androgen withdrawal).
* Rising serum PSA (Prostate Cancer Working Group (PCWG2) definition).
* Castrate levels of serum testosterone (i.e., ≤ 50 ng/dL).
* Age > 18 years.
* ECOG performance status score ≤ 2, and/or Karnofsky score ≥ 50%.
* Life expectancy > 6 months.
* Adequate kidney, liver, and bone marrow function.
* Willingness to sign informed consent and adhere to study requirements.

Exclusion Criteria:

* Recent surgery, radiation therapy, combined androgen blockade, or investigational therapies in the last 8 weeks.
* Previous chemotherapy for metastatic prostate cancer.
* Concomitant use of second-line hormonal agents (e.g., ketoconazole, DES)
* Current use of corticosteroids, except if on a stable dose for ≥ 3 months.
* History of malabsorption syndrome (may affect itraconazole absorption).
* Allergic reactions to itraconazole or similar compounds.
* Concurrent use of drugs that interact with the CYP3A4 system (caution only).
* Presence of known brain metastases.
* Prior malignancy in the last 3 years, with some exceptions.
* Uncontrolled major infectious, cardiac, or pulmonary illnesses.
* Prolonged corrected QT interval (> 450 msec) on electrocardiography.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-07; Primary Completion 2011-05 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Carducci, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose | High Dose
Started | 17 | 29
Completed | 17 | 25
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose | High Dose | Total
Number analyzed (Participants) | 17 | 29 | 46
Age, Continuous [Median (Full Range); unit: years] | 73 [60 to 81] | 71 [52 to 89] | 73 [52 to 89]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 9 | 10
  >=65 years | 16 | 20 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 29 | 46
Region of Enrollment [Number; unit: participants]
  United States | 17 | 29 | 46

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Proportion of Patients With Metastatic CRPC Who do Not Have Prostate Specific Antigen (PSA) Progression After 24 Weeks of Therapy With One of Two Dose-levels of Itraconazole: 200 mg or 600 mg Daily.
Description: To Determine the Proportion of Patients With Metastatic CRPC Who do Not Have Prostate Specific Antigen (PSA) Progression After 24 Weeks of Therapy. "PSA progression" is defined as a 25% increase in PSA over baseline [or nadir (lowest)] and an increase in absolute PSA level by at least 2 ng/mL, both confirmed by a second value at least 4 weeks later.
Time Frame: Up to 24 weeks
Population: Based on how many participants were evaluable for the study primary endpoint
Measure: Number (95% Confidence Interval); unit: percent of patients
Groups:
- Low Dose Itraconazole: Itraconazole, 200 mg, by mouth, once daily (200 mg total daily dose)
  Itraconazole 200 mg: Itraconazole, 200 mg, by mouth, once daily (200 mg total daily dose)
- High Dose Itraconazole: Itraconazole, 300 mg, by mouth, twice daily (600 mg total daily dose)
  Itraconazole 300mg: Itraconazole, 300 mg, by mouth, twice daily (600 mg total daily dose)
Arm/Group | Low Dose Itraconazole | High Dose Itraconazole
Number analyzed (Participants) | 17 | 25
percent of patients | 11.8 [1.5 to 36.4] | 48 [27.8 to 68.7]

2. Secondary Outcome: To Determine the Proportion of Men With ≥ 50% PSA Reduction From Baseline.
Description: Will be reported as the percentage of men with ≥ 50% PSA reduction from baseline.
Time Frame: Baseline and approximately 2 years from open enrollment
Population: One subject in the high dose arm was not evaluable on account of subject discontinuing study drug during cycle 1 due to clinical progression.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Low Dose | High Dose
Number analyzed (Participants) | 17 | 28
percentage | 0 [0 to 19.5] | 14.3 [4.0 to 32.7]

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Low Dose | High Dose
Serious Adverse Events (participants affected / at risk) | 1/17 | 0/29
Other Adverse Events (participants affected / at risk) | 14/17 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=17) | High Dose (N=29)
fatigue (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=17) | High Dose (N=29)
fatigue (General disorders) | 9 (9) | 6 (6)
anorexia (Gastrointestinal disorders) | 2 (2) | 5 (5)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
hypertension (Cardiac disorders) | 0 (0) | 9 (9)
hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes